CLINICAL TRIAL: NCT05043337
Title: The Effects of the Maternal Voice Combined With Lullaby to Reduce the Heel Puncture Pain in Preterm Infant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Y_110_0206
Record Dates: First submitted 2021-09-05; First posted 2021-09-14 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Pain
Keywords: premature; maternal voice; lullaby; heel punture; neonatal pain
MeSH Terms: conditions — Pain; Premature Birth

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Maternal voice (Experimental): Recording the maternal voice in reading children's books, and recorded the sound for 13 minutes. When the premature infants undergoing heel lance procedure, the experimental group was explored maternal voice, which starts from 3 minutes before the procedure and ends ten minutes after the heel puncture.
  Interventions: Behavioral: Maternal voice
- Lullaby (Experimental): The Brahms Lullaby recordings are compiled for 13 minutes. When the premature infants undergoing heel lance procedure, the experimental group was explored Brahms Lullaby, which starts from 3 minutes before the procedure and ends ten minutes after the heel puncture.
  Interventions: Behavioral: Lullaby
- Maternal voice combined with lullaby (Experimental): Recording the maternal voice in reading children's books and giving mother listening to the lullaby at the same time, and recorded the sound for 13 minutes. When the premature infants undergoing heel lance procedure, the experimental group was explored Maternal voice combined with Brahms lullaby, which starts from 3 minutes before the procedure and ends ten minutes after the heel puncture.
  Interventions: Behavioral: Maternal voice combined with lullaby
- Control group (No Intervention): When the premature infants undergoing heel lance procedure , the control group was under routine care . Measuring with the Respiration , heart rate , oxygen saturation , and neonatal infant pain scale (NIPS ) were recorded 3 minutes before , during , 1st , 3rd , and 10th minutes after the heel lance puncture .

INTERVENTIONS:
Behavioral: Maternal voice — The recordings were made in a quiet and separate consultation room. For infants in the "maternal voice group," mothers were recorded what they wanted to say to their baby and read an independently published children's book, "Xiao Qi's yellow persimmon" which describes how mothers with premature babies care for their infants. After reviewing the quality of the recordings, the maternal voice recordings were edited for 13 minutes using a sound organizer. Respiration, heart rate, oxygen saturation, and Neonatal Infant Pain Scale (NIPS) were measured and recorded 3 minutes before, during, 1 minute, 3 minutes, and 10 minutes after the puncture.
  Arms: Maternal voice
Behavioral: Lullaby — The Brahms Lullaby recordings are compiled for 13 minutes. Measuring with the Respiration, heart rate, oxygen saturation, and neonatal infant pain scale (NIPS ) were recorded 3 minutes before, during, 1st, 3rd, and 10th minutes after the heel lance puncture.
  Arms: Lullaby
Behavioral: Maternal voice combined with lullaby — The recordings were made in a quiet and separate consultation room. For infants in the " Maternal voice combined with lullaby group, " mothers were recorded what they wanted to say to their baby and read an independently published children's book-"Xiao Qi's yellow persimmon ", and giving mother listening to the Brahms Lullaby at the same time, the maternal voice recordings were edited for 13 minutes using a sound organizer. Measuring with the Respiration, heart rate, oxygen saturation, and neonatal infant pain scale (NIPS ) were recorded 3 minutes before, during, 1st, 3rd, and 10th minutes after the heel lance puncture.
  Arms: Maternal voice combined with lullaby

SUMMARY:
In Taiwan, 183,254 newborns were born in 2018, with preterm births accounting for about 8-10%. The preterm infant required frequent medical treatment from birth to hospital discharge, which is accompanied by a painful process that can cause unstable vital signs in the short term and may affect their biological and psychological development in the long term. Music therapy is a non-invasive and easily accessible intervention, can be used to reduce the discomfort of painful stimulation during hospitalization of preterm infants. Music therapies in this text are the mother's voice and lullabies.

DETAILED DESCRIPTION:
This study was a quantitative study of a randomized controlled trial, designed by experimental research method, and followed the principle of Allocation Concealment to conduct a randomized assignment trial. Using G*Power 3.1 to estimate the number of samples, and the statistical method chosen was Repeated measures ANOVA, the sample size is 120.

The subjects were divided into four groups, all four groups were administered general routine care, three experimental groups, and one control group, and the experimental group was a repetitive segment of audio recording edited to 13 minutes. There were three interventions: group A maternal voice reading children's books, group B lullaby, group C maternal voice reading children's books combined with lullaby, and the control group was the routine care group without any audio intervention. Physiological indicators, including heart rate, respiratory rate, oxygen saturation, and pain response assessed using the Neonatal Infant Pain Scale (NIPS), were recorded 3 minutes before, during, 1st, 3rd, and 10 minutes after heel lance puncture.

ELIGIBILITY:
Inclusion Criteria:

1. Babies born alive before 37 weeks of pregnancy.
2. Infants who were required to receive heel lance procedure every 8 hours after physicians' diagnoses.
3. Those who can record the mother's voice and whose mother can read Chinese.

Exclusion Criteria:

1. Abnormal ear appearance, chromosomal abnormalities, congenital or acquired infections.
2. Postnatal patients whose mothers are not in the postnatal ward, e.g., those who need to be admitted to the intensive care unit due to their medical condition.
3. Patients used high-frequency oscillatory ventilators, because the high-frequency oscillatory ventilator gives 600 oscillatory breaths per minute and it is not possible to evaluate whether the study subjects can effectively listen to the interventions given, so they were excluded.
4. Mothers who were unable to complete the recording because of emotional ups and downs during the recording process.
5. Mothers who smoked, drank alcohol or used illegal drugs during pregnancy.
6. the patients was diagnosed with Asphyxia of the newborn at birth
7. Painkillers used within 2 days of birth.

Ages: 2 Days to 2 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2021-10-31 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-02-06 (Actual)

PRIMARY OUTCOMES:
Heart rate | Change from Baseline Heart rate at 3 minutes before, during, and at 1st、3rd and 10th minute after heel lance procedure
  Using the German-made PHILIPS IntelliVue MP40 Dräger Julian physiological index monitor, including monitoring Heart Rate (HR).
Respiratory rate | Change from Baseline Respiratory rate at 3 minutes before, during, and at 1st、3rd and 10th minute after heel lance procedure
  Using the German-made PHILIPS IntelliVue MP40 Dräger Julian physiological index monitor, including monitoring Respiratory rate (RR).
Oxygen Saturation | Change from Baseline Saturation of Peripheral Oxygen at 3 minutes before, during, and at 1st、3rd and 10th minute after heel lance procedure
  Using the German-made PHILIPS IntelliVue MP40 Dräger Julian physiological index monitor, including monitoring Saturation of Peripheral Oxygen (SPO2).
Respond of Pain | Change from Baseline Pain at 3 minutes before, during, and at 1st、3rd and 10th minute after heel lance procedure
  Pain response assessed using the Neonatal Infants Pain Scale (NIPS), The evaluation indicators include 6 behavior indicators: facial expression, crying, breathing pattern, arms, legs, and awakening status, except that the crying score is divided into three points (0, 1, 2 points), and the rest are two points (0 , 1 point), the total score is 0-7 points, the higher the score, the more serious the pain.

CONTACTS AND LOCATIONS:
Locations (1):
- National Yang Ming Chiao Tung University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Filippa M, Panza C, Ferrari F, Frassoldati R, Kuhn P, Balduzzi S, D'Amico R. Systematic review of maternal voice interventions demonstrates increased stability in preterm infants. Acta Paediatr. 2017 Aug;106(8):1220-1229. doi: 10.1111/apa.13832. Epub 2017 Apr 19. PMID 28378337
- [Background] Chirico G, Cabano R, Villa G, Bigogno A, Ardesi M, Dioni E. Randomised study showed that recorded maternal voices reduced pain in preterm infants undergoing heel lance procedures in a neonatal intensive care unit. Acta Paediatr. 2017 Oct;106(10):1564-1568. doi: 10.1111/apa.13944. Epub 2017 Jul 5. PMID 28580602
- [Background] Polkki T, Korhonen A. The effectiveness of music on pain among preterm infants in the neonatal intensive care unit: a systematic review. JBI Libr Syst Rev. 2012;10(58):4600-4609. doi: 10.11124/jbisrir-2012-428. PMID 27820525
- [Background] Jabraeili M, Sabet T, MustafaGharebaghi M, Asghari Jafarabadi M, Arshadi M. The Effect of Recorded Mum's Lullaby and Brahm's Lullaby on Oxygen Saturation in Preterm Infants: a Randomized Double-Blind Clinical Trial. J Caring Sci. 2016 Mar 1;5(1):85-93. doi: 10.15171/jcs.2016.009. eCollection 2016 Mar. PMID 26989669
- [Background] Uematsu H, Sobue I. Erratum: Effect of music (Brahms lullaby) and non-nutritive sucking on heel lance in preterm infants: A randomized controlled crossover trial. Paediatr Child Health. 2019 Feb;24(1):63. doi: 10.1093/pch/pxy163. Epub 2018 Dec 14. PMID 30793710